CLINICAL TRIAL: NCT04435067
Title: Retrospective Observational Study on Patients With Lung Metastases From Pancreatic Adenocarcinoma: Evaluation of Clinical Features and Correlation With Molecular and Radiomics Features
Brief Title: Evaluation of Clinical, Radiomics and Molecular Features of Lung Metastasis in PDAC Patients (LUMACA Trial)
Acronym: LUMACA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Michele Reni, MD, IRCCS San Raffaele
Other Study IDs: PACT32
Record Dates: First submitted 2020-06-14; First posted 2020-06-17 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Pancreas Adenocarcinoma
Keywords: Pancreas Adenocarcinoma; Lung Metastasis; Gene Expression; Molecular analysis; Radiomics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — DNA from histological samples fixed in formalin and included in paraffin
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort A: patients in whom lung metastasis were resected for therapeutic purposes
  Interventions: Genetic: Analysis of genetic mutations and the gene expression profile of lung metastasis and primary neoplasia; Other: Radiomics analysis on TAC imaging at diagnosis of lung metastasis and, if possible, of the primary tumor
- Cohort B: patients in whom lung metastasis were removed for diagnostic purposes only
  Interventions: Genetic: Analysis of genetic mutations and the gene expression profile of lung metastasis and primary neoplasia; Other: Radiomics analysis on TAC imaging at diagnosis of lung metastasis and, if possible, of the primary tumor

INTERVENTIONS:
Genetic: Analysis of genetic mutations and the gene expression profile of lung metastasis and primary neoplasia — The mutational analysis of the main oncogenes and tumor suppressor genes involved in the genesis and tumor progression will be performed on the genomic DNA extracted from each sample using the Ion Torrent TM Oncomine TM Comprehensive Assay version 3 (OCAv3) kit. This panel includes 161 cancer-related genes and allows the identification of all genomic alterations affecting oncogenes and recurrently altered tumor suppressor genes in solid tumors. The study of gene expression will be carried out using Nanostring Technology using the Pancancer IO 360 TM panel which allows simultaneous analysis for each sample of multiple mRNAs associated with crucial pathways in carcinogenesis and the immunological profile of the tumor, defining its up and down conditions gene regulation.
Other: Radiomics analysis on TAC imaging at diagnosis of lung metastasis and, if possible, of the primary tumor — This study will be performed using the SPAARC IBSI (International Biomarker Standardization Initiative) compliant software implemented in the MatLab environment (MathWorks, Boston, USA) through several steps: (a) CT imaging retrieval, (b) image segmentation and rendering, (c) feature extraction and (d) qualification/quantification. Approximately 200 radiomics characteristics will be extracted, such as: Morphology, Statistical, Intensity Histogram, Gray Level Co-occurrence Matrix 3D_average, Gray Level Co-occurrence Matrix 3D_combined, Gray Level Run Length 3D_average, Gray Level Run Length 3D_combined, Gray Level Size Zone Matrix 3D, Neighbor Gray Tone Difference Matrix 3D, Gray Level Distance Zone Matrix 3D.

SUMMARY:
The aim of this study is the characterization from epidemiological, radiomics and molecular point of view of lung metastasis of patients at beginning affected by pancreatic adenocarcinoma (PDAC), which after the resection of primitive tumor have met with initial recurrence of the disease exclusively at the lung level.

DETAILED DESCRIPTION:
Radical surgical treatment of primitive PDAC, associated with adjuvant cancer treatments, is possible only in 15-20% of patients, and, to date, represents the best therapeutic strategy. Nevertheless, remote recurrence is frequent after radical surgical treatment of primitive neoplasia. Among the main locations of metastasis from PDAC, the lung represent the second metastatic location with a better prognosis than other remote metastasis. Surgical treatment of lung metastasis has a consolidated role in the treatment of other neoplasms such as sarcomas, colorectal and renal neoplasms while in the context of PDAC the resection of lung metastases is a rather rare and also debated event.

In absence of consolidated data on the results of surgical treatment and on the clinical outcomes of patients with lung metastasis from PDAC the investigators designed this retrospective observational study in order to analyze the clinical and pathological characteristics of patients suffering from lung metastasis from PDAC treated at San Raffaele Hospital in a period between 2008 and 2019. To this purpose, the investigators will analyze and compare two patient cohorts: 1-patients in whom lung metastasis were resected for therapeutic purposes; 2-patients in whom lung metastasis were removed for diagnostic purposes only.

An analysis of genetic mutations and the gene expression profile of lung metastasis and primary neoplasia will also be performed to evaluate any predictive elements of lung metastasis and the prognostic role of these mutations.

In parallel, the investigators will perform radiomics analysis on TAC imaging at diagnosis of lung metastasis and, if possible, of the primary tumor.

All the data necessary for the completion of the study were collected as part of the usual outpatient visits in the appropriate outpatient medical records and include: date of birth, date of diagnosis, gender, performance status, stage of the disease, comorbidity, concomitant chronic therapies, level of tumor markers (CEA and Ca19.9) before treatment and variations during therapy, type of chemotherapy, start and end date of chemotherapy, number of cycles, possible dosage reduction of the drugs used in the various chemotherapy regimes, dates and results of instrumental revaluations according to RECIST 1.1, main chemotherapy toxicities and grade according to CTCAE 5.0, date and type of surgery, mutation analysis results and last follow-up date. In the event of death, the dates of death are communicated by the registry office of the municipality of residence of the patient, according to the official procedure. All data will be collected in an electronic database in coded form (pseudonymization).

Power size calculation:

All patients who meet the inclusion and exclusion criteria and who have been treated at the Medical Oncology and Thoracic Surgery Units of the San Raffaele Hospital between 2008 and 2019 will be taken into consideration, for a total of 44 patients. To identify predictive and/or prognostic clinical and pathological factors that can influence the outcome of these patients, the two cohorts described above will be analyzed and compared through univariate and multivariate analyzes. Overall survival (OS) and progression-free survival (PFS) will also be assessed using the Kaplan Meier method and the long-rank test will be used to compare OS and PFS between the two cohorts under study. All tests will be double-tailed and a p <0.05 will be considered significant. The ninety-five percent confidence intervals (CI) will be calculated to assess the accuracy of the estimates obtained.

ELIGIBILITY:
Inclusion Criteria:

* Cytological/histological diagnosis of pancreatic adenocarcinoma as a primary tumor and localization of adenocarcinoma compatible with pancreatic primitivity for lung metastasis;
* Previous surgical resection of the primary tumor;
* Exclusive presence of single or multiple lung metastasis at disease recurrence;
* Radical or diagnostic excision of lung metastasis;
* Informed patient consent (for currently living patients).

Exclusion Criteria:

* Patients not undergoing lung resection surgery for diagnostic and/or therapeutic purposes for cardiac or respiratory functional contraindication.
* Patients with lung metastases synchronous with primary cancer. Contacts and Locations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with a confirmed diagnosis of lung metastasis from PDAC from 2008 to 2019
Sampling Method: Non-Probability Sample
Enrollment: 44 (Estimated)
Dates: Start 2020-05-27 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical and pathological features of lung metastasis | 6 months
  Analyze the clinical and pathological characteristics of the two cohorts of patients affected by lung metastasis from PDAC

SECONDARY OUTCOMES:
Molecular and radiomics features of lung metastasis | 18 months
  Correlate the pathological characteristics of the two cohorts of patients affected by lung metastasis from PDAC with radiomics and molecular features, in order to identify prognostic and/or predictive factors related to lung metastasis in the PDAC
Differences between the two cohorts | 18 months
  Highlight any differences between the two cohorts of patients examined

CONTACTS AND LOCATIONS:
Overall Officials: Michele Reni, MD, Principal Investigator — IRCCSS Raffaele
Locations (4):
- Italy (4):
  - IRCCS San Raffaele Diagnostic Radiology Unit, Milan
  - IRCCS San Raffaele Medical Oncology Unit, Milan
  - IRCCS San Raffaele Pathological Anatomy Unit, Milan
  - IRCCS San Raffaele Thoracic Surgery Unit, Milan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arnaoutakis GJ, Rangachari D, Laheru DA, Iacobuzio-Donahue CA, Hruban RH, Herman JM, Edil BH, Pawlik TM, Schulick RD, Cameron JL, Meneshian A, Yang SC, Wolfgang CL. Pulmonary resection for isolated pancreatic adenocarcinoma metastasis: an analysis of outcomes and survival. J Gastrointest Surg. 2011 Sep;15(9):1611-7. doi: 10.1007/s11605-011-1605-8. Epub 2011 Jul 2. PMID 21725701
- [Background] Ceppa DP. Results of Pulmonary Resection: Sarcoma and Germ Cell Tumors. Thorac Surg Clin. 2016 Feb;26(1):49-54. doi: 10.1016/j.thorsurg.2015.09.007. PMID 26611510
- [Background] Okui M, Yamamichi T, Asakawa A, Harada M, Horio H. Resection for Pancreatic Cancer Lung Metastases. Korean J Thorac Cardiovasc Surg. 2017 Oct;50(5):326-328. doi: 10.5090/kjtcs.2017.50.5.326. Epub 2017 Oct 5. PMID 29124023
- [Background] Rama N, Monteiro A, Bernardo JE, Eugenio L, Antunes MJ. Lung metastases from colorectal cancer: surgical resection and prognostic factors. Eur J Cardiothorac Surg. 2009 Mar;35(3):444-9. doi: 10.1016/j.ejcts.2008.10.047. Epub 2009 Jan 10. PMID 19136273
- [Background] Yamashita K, Miyamoto A, Hama N, Asaoka T, Maeda S, Omiya H, Takami K, Doki Y, Mori M, Nakamori S. Survival Impact of Pulmonary Metastasis as Recurrence of Pancreatic Ductal Adenocarcinoma. Dig Surg. 2015;32(6):464-71. doi: 10.1159/000439545. Epub 2015 Oct 31. PMID 26517228